CLINICAL TRIAL: NCT00696215
Title: The Effects of Rasagiline on Cognitive Deficits Associated With Parkinson's Disease: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study Over 3 Months
Brief Title: The Effects of Rasagiline on Cognitive Deficits Associated With Parkinson's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Prof. Murat Emre, Istanbul Faculty of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11719A
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; rasagiline; cognition; MAO-B
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Active Comparator): Rasagiline
  Interventions: Drug: rasagiline

INTERVENTIONS:
Drug: placebo — Placebo 1 mg once a day
  Arms: 1
Drug: rasagiline — 1mg
  Other Names: Azilect
  Arms: 2

SUMMARY:
The objective of the study is to assess the effects of rasagiline on cognitive functions in patient with Parkinson's disease. Patients on any dopaminergic medications will be assigned to receive rasagiline 1 mg or placebo over 3 months. Cognitive functions will be assessed by selected neuropsychological tests representing each cognitive domain.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the effects of rasagiline on cognitive deficits in non-demented patients with PD. The secondary objective is to assess affective changes in this patient population. This will be a randomized, double-blind, placebo controlled study in 1-3 centers. Patients will be recruited from the Movement Disorders Outpatients Clinic, Department of Neurology, Istanbul Faculty of Medicine, Dokuz Eylul University and Marmara University. Eligible patients will be randomly assigned to rasagiline 1 mg or placebo. Patients will be treated with the study medication over 3 months. Cognitive and behavioral assessments will be performed at baseline, at 4 weeks and at the end of the study, at 12 weeks. A total of 40 PD patients with cognitive deficits, but without dementia will be recruited. No sample size calculation will be performed, a sample of convenience will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients of any age
2. Diagnosis of Idiopathic PD according to the UK Brain Bank Criteria for the clinical diagnosis of PD.
3. Patients with cognitive impairment associated with PD, defined as:

   1. Subjective complaints of impaired cognitive functions such as forgetfulness, word finding difficulties or inattentiveness
   2. Presence of objectively demonstrable cognitive deficits in at least 2 out of the 4 cognitive domains typically impaired in PD. These include attention, executive functions, memory and visuo-spatial functions. The performance in the following test scores must be 1.5 standard deviations below the mean normative score for age and education of the patient: Digit Span for attention, Letter Fluency test for executive function, Logical Memory Sub-scale from the Wechsler Memory Scale-Revised and Line Orientation Test for visuo-spatial function.
4. Patients with a Hoehn and Yahr stage I-III when "on"
5. Literate patients who are able to follow test instructions

Exclusion Criteria:

1. Diagnosis of dementia due to PD according to DSM IV criteria
2. Diagnosis of current major depressive episode according to DSM IV criteria
3. Presence of any other neurodegenerative disorder other than PD
4. Presence of any unstable or untreated systemic disorder such as diabetes, cardiac failure, renal failure
5. Use of any prohibited concomitant medication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-06 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will be the total cognitive score. This will be calculated by adding the four cognitive sub-scores: attention, executive function, memory and visuo-spatial function. | 30 months

SECONDARY OUTCOMES:
The four cognitive sub-scores as well as individual tests scores will be analyzed separately. The changes from baseline to the end of the study in the GDS, STAS and UPDRS part III scales will be analyzed. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: MURAT EMRE, PROF, Principal Investigator — ISTANBUL FACULTY OF MEDICINE
Locations (2):
- Turkey (Türkiye) (2):
  - Marmara University, Istanbul
  - Raif Cakmur, Izmir